CLINICAL TRIAL: NCT02226822
Title: J-DISCOVER: DISCOVERing Treatment Reality of Type 2 Diabetes in Real World Setting in Japan
Brief Title: DISCOVERing Treatment Reality of Type 2 Diabetes in Real World Setting in Japan
Acronym: J-DISCOVER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D1692R00001
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients with documented T2DM: Adult patients with documented history of type 2 diabetes mellitus who are initiating their second line oral or parenteral anti-diabetics medication after first line oral diabetic therapy

SUMMARY:
This study is intended to prospectively research the treatment reality and long-term disease control of Type 2 Diabetes Mellitus (T2DM) patients who are initiating 2nd line anti-diabetes treatment in sites across Japan.

DETAILED DESCRIPTION:
This study is a single country, multicenter, observational, prospective, longitudinal cohort study which will include adult patients with documented history of T2DM who are initiating a second line oral or parenteral anti-diabetes mediation after their first line anti-diabetic therapy in real world setting. The follow-up period is 3 years. Patients will undergo clinical assessments and receive standard medical care as determined by the treating physician. Patients will not receive experimental intervention or experimental treatment as a consequence of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent obtained
2. Aged > = 20 years
3. Diagnosed with type 2 diabetes mellitus
4. Initiating a second oral or parenteral anti-diabetic therapy added to oral anti-diabetic monotherapy or switching from the monotherapy to another monotherapy with different drug class

Exclusion Criteria:

1. Diagnosis of Type 1 Diabetes Mellitus
2. Current pregnancy
3. Current treatment for any cancer
4. Current dialysis treatment or renal transplantation
5. Current treatment with any oral steroids
6. Participation in any randomized control trials
7. Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker who does not understand the local language where interpreter are not available, psychiatric disturbances, alcohol or drug abuse).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with documented history of type 2 diabetes mellitus who are initiating their second line oral or parenteral anti-diabetics medication after first line oral diabetic therapy
Sampling Method: Non-Probability Sample
Enrollment: 1869 (Actual)
Dates: Start 2014-09-20 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Classes of diabetic medications at baseline and changes up to 3 years | At 6, 12, 24, 36 month from enrollment
  Classes of anti-diabetic medications at baseline and any changes of anti-diabetic medications during 3 years follow-up period.

SECONDARY OUTCOMES:
Hemoglobin A1c change from baseline, Achievement rate of HbA1c and blood glucose target goals | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, treatment response in terms of changes in HbA1c from baseline, achievement rate of HbA1c and blood glucose target goals
Blood glucose level change from baseline | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, treatment response in terms of changes in blood glucose level (FPG or CPG or PPG) from baseline.
Body weight change from baseline | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, treatment response in terms of changes in body weight.
Blood pressure change from baseline | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, treatment response in terms of changes in blood pressure from baseline.
Lipid profile changes from baseline | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, treatment response in terms of changes in lipid profile
Incidence of microvascular complications | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, disease progression in terms of microvascular complications: incidence of chronic nephropathy, dialysis, diabetic retinopathy, retinal photocoagulation, amputation of lower extremity, diabetic foot, peripheral nerve disorders, autonomic nervous system disorders and erectile dysfunction.
Hypoglycemia events | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, hypoglycemic events and hyperglycermia hospitalizations
Patient reported Quality of Life, diet, and physical activity level | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, patient reported Quality of Life, diet, and physical activity level
Initiation of insulin therapy, Proportion of patients using insulin | At 6, 12, 24, 36 month from enrollment
  Initiation of insulin therapy (e.g., reporting the average number of anti-diabetic therapies prescribed as insulin therapy is initiated and dose of insulin)
Switching of anti-diabetic medications or dose change | At 6, 12, 24, 36 month from enrollment
  Switching of anti-diabetic medications or dose change
Initiation of third line or above add-on anti-diabetic medications | At 6, 12, 24, 36 month from enrollment
  Initiation of third line or above add-on anti-diabetic medication (e.g., reporting proportion of patients receiving 2nd, 3rd, 4th or greater anti-diabetic therapies at each follow-up visit)
Incidence of macrovascular complications | At 6, 12, 24, 36 month from enrollment
  Overall and by second line anti-diabetic medication class, disease progression in terms of macrovascular complications (heart failure, myocardial infarction and stroke).
Risk factors | At 6, 12, 24, 36 month after enrollment
  Risk factors (patient characteristics at baseline: e.g. age, gender, duration of diabetes, presence of co-morbidities) associated with poorer clinical outcomes during follow-up
Treatment choice | At baseline
  Determinants of treatment choice

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Hashigami, M.D., Study Director — AstraZeneca; Iichiro Shimomura, M.D., Ph.D., Principal Investigator — Department of Metabolic Medicine (Internal Medicine), Graduate School of Medicine, Osaka University; Hirotaka Watada, M.D., Ph.D., Principal Investigator — Department of Metabolism & Endocrinology, Graduate School of Medicine, Juntendo University
Locations (106):
- Japan (106):
  - Research Site, Anjo, Aichi-ken
  - Research Site, Anzai, Aichi-ken
  - Research Site, Komatsu, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Hirosaki, Aomori
  - Research Site, Funabashi, Chiba
  - Research Site, Kisarazu, Chiba
  - Research Site, Tateyama, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Ono, Fukui
  - Research Site, Itoshima, Fukuoka
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Kurate-gun, Fukuoka
  - Research Site, Oguri, Fukuoka
  - Research Site, Ōnojō, Fukuoka
  - Research Site, Iwaki, Fukushima
  - Research Site, Shirakawa, Fukushima
  - Research Site, Isesaki, Gunma
  - Research Site, Kanra-gun, Gunma
  - Research Site, Shibukawa, Gunma
  - Research Site, Takasaki, Gunma
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Hakodate, Hokkaido
  - Research Site, Kamikawa, Hokkaido
  - Research Site, Muroran, Hokkaido
  - Research Site, Nakagawa, Hokkaido
  - Research Site, Otaru, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Amagasaki, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Tamba, Hyōgo
  - Research Site, Hitachi, Ibaraki
  - Research Site, Koga, Ibaraki
  - Research Site, Ushiku, Ibaraki
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Komatsu, Ishikawa-ken
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Kanoya, Kagoshima-ken
  - Research Site, Chigasaki, Kanagawa
  - Research Site, Hiratsuka, Kanagawa
  - Research Site, Isehara, Kanagawa
  - Research Site, Kamakura, Kanagawa
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Hitoyoshi, Kumamoto
  - Research Site, Tamana, Kumamoto
  - Research Site, Ise, Mie-ken
  - Research Site, Tsu, Mie-ken
  - Research Site, Yokkaichi, Mie-ken
  - Research Site, Sendai, Miyagi
  - Research Site, Nichinan, Miyazaki
  - Research Site, Iida, Nagano
  - Research Site, Ueda, Nagano
  - Research Site, Kitakatsuragi-gun, Nara
  - Research Site, Jōetsu, Niigata
  - Research Site, Tomigusuku, Okinawa
  - Research Site, Urazoe, Okinawa
  - Research Site, Ikuno-ku, Osaka
  - Research Site, Kashihara, Osaka
  - Research Site, Sennan-gun, Osaka
  - Research Site, Toyonaka, Osaka
  - Research Site, Imari, Saga-ken
  - Research Site, Karatsu, Saga-ken
  - Research Site, Nishimatuura, Saga-ken
  - Research Site, Kasukabe, Saitama
  - Research Site, Sakado, Saitama
  - Research Site, Kouka, Shiga
  - Research Site, Kōka, Shiga
  - Research Site, Maibara, Shiga
  - Research Site, Ōtsu, Shiga
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Yaizu, Shizuoka
  - Research Site, Nasushiobara, Tochigi
  - Research Site, Oyama, Tochigi
  - Research Site, Shimotsuga-gun, Tochigi
  - Research Site, Edogawa-ku, Tokyo
  - Research Site, Hachiōji, Tokyo
  - Research Site, Kita-ku, Tokyo
  - Research Site, Koganei, Tokyo
  - Research Site, Kokubunji, Tokyo
  - Research Site, Mitaka, Tokyo
  - Research Site, Nerima-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Iwade, Wakayama
  - Research Site, Nakami, Yamagata
  - Research Site, Ube, Yamaguchi
  - Research Site, Kofu, Yamanashi
  - Research Site, Chiba
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Hiroshima
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Miyazaki
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Yamagata

REFERENCES:
- [Derived] Al Rubeaan K, Banah F, Alruwaily FG, Sheshah E, Alnaqeb D, AlQahtani AM, Ewais D, Al Juhani N, Hassan AH, Youssef AM. Metabolic control and incidence of hypoglycaemia, hospitalisation and complications among Saudi patients with type 2 diabetes initiating second-line therapy: an analysis of the Saudi Arabia data from the DISCOVER Observational Study programme. BMJ Open. 2023 Aug 30;13(8):e063586. doi: 10.1136/bmjopen-2022-063586. PMID 37648382
- [Derived] Mita T, Katakami N, Takahara M, Kawashima M, Wada F, Akiyama H, Morita N, Kidani Y, Yajima T, Shimomura I, Watada H. Changes in Treatment Satisfaction Over 3 Years in Patients With Type 2 Diabetes After Initiating Second-line Treatment. J Clin Endocrinol Metab. 2022 Aug 18;107(9):2424-2432. doi: 10.1210/clinem/dgac420. PMID 35857060
- [Derived] Hejjaji V, Gorgojo-Martinez JJ, Tang F, Garnelo JB, Cooper A, Medina J, Mutiozabal MS, Khunti K, Nicolucci A, Shestakova MV, Ji L, Gomes MB, Watada H, Vora J, Malik AO, Kosiborod M, Arnold SV. Factors associated with weight loss in people with overweight or obesity living with type 2 diabetes mellitus: Insights from the global DISCOVER study. Diabetes Obes Metab. 2022 Sep;24(9):1734-1740. doi: 10.1111/dom.14745. Epub 2022 May 25. PMID 35546275
- [Derived] Takahara M, Mita T, Katakami N, Wada F, Morita N, Kidani Y, Yajima T, Shimomura I, Watada H; J-DISCOVER study group. Three-Year Glycaemic Control and Management in Patients with Type 2 Diabetes Initiating Second-Line Treatment in Japan: A Prospective Observational Study, J-DISCOVER. Diabetes Ther. 2022 Feb;13(2):251-264. doi: 10.1007/s13300-021-01192-x. Epub 2021 Dec 28. PMID 34962628
- [Derived] Khunti K, Gomes MB, Kosiborod M, Nicolucci A, Pocock S, Rathmann W, Shestakova MV, Shimomura I, Watada H, Chen H, Cid-Ruzafa J, Fenici P, Hammar N, Tang F, Ji L; DISCOVER Scientific Committee and all DISCOVER investigators. Metformin discontinuation in patients beginning second-line glucose-lowering therapy: results from the global observational DISCOVER study programme. BMJ Open. 2020 Aug 30;10(8):e034613. doi: 10.1136/bmjopen-2019-034613. PMID 32868349
- [Derived] Katakami N, Mita T, Takahara M, Yajima T, Wada F, Kawashima M, Shimomura I, Watada H; J-DISCOVER Study Group. Baseline Characteristics of Patients with Type 2 Diabetes Initiating Second-Line Treatment in Japan: Findings from the J-DISCOVER Study. Diabetes Ther. 2020 Jul;11(7):1563-1578. doi: 10.1007/s13300-020-00846-6. Epub 2020 Jun 5. PMID 32504219
- [Derived] Khunti K, Chen H, Cid-Ruzafa J, Fenici P, Gomes MB, Hammar N, Ji L, Kosiborod M, Pocock S, Shestakova MV, Shimomura I, Tang F, Watada H, Nicolucci A; DISCOVER investigators. Glycaemic control in patients with type 2 diabetes initiating second-line therapy: Results from the global DISCOVER study programme. Diabetes Obes Metab. 2020 Jan;22(1):66-78. doi: 10.1111/dom.13866. Epub 2019 Oct 1. PMID 31468637
- [Derived] Nicolucci A, Charbonnel B, Gomes MB, Khunti K, Kosiborod M, Shestakova MV, Shimomura I, Watada H, Chen H, Cid-Ruzafa J, Fenici P, Hammar N, Surmont F, Tang F, Pocock S. Treatment patterns and associated factors in 14 668 people with type 2 diabetes initiating a second-line therapy: Results from the global DISCOVER study programme. Diabetes Obes Metab. 2019 Nov;21(11):2474-2485. doi: 10.1111/dom.13830. Epub 2019 Aug 5. PMID 31297947
- [Derived] Khunti K, Ji L, Medina J, Surmont F, Kosiborod M. Type 2 diabetes treatment and outcomes worldwide: A short review of the DISCOVER study programme. Diabetes Obes Metab. 2019 Nov;21(11):2349-2353. doi: 10.1111/dom.13817. Epub 2019 Jul 14. PMID 31215715
- [Derived] Kosiborod M, Gomes MB, Nicolucci A, Pocock S, Rathmann W, Shestakova MV, Watada H, Shimomura I, Chen H, Cid-Ruzafa J, Fenici P, Hammar N, Surmont F, Tang F, Khunti K; DISCOVER investigators. Vascular complications in patients with type 2 diabetes: prevalence and associated factors in 38 countries (the DISCOVER study program). Cardiovasc Diabetol. 2018 Nov 28;17(1):150. doi: 10.1186/s12933-018-0787-8. PMID 30486889
- [Derived] Katakami N, Mita T, Takahara M, Hashigami K, Kawashima M, Shimomura I, Watada H; J-DISCOVER study group. Rationale and Design for the J-DISCOVER Study: DISCOVERing the Treatment Reality of Type 2 Diabetes in a Real-World Setting in Japan-A Protocol. Diabetes Ther. 2018 Feb;9(1):165-175. doi: 10.1007/s13300-017-0351-7. Epub 2017 Dec 19. PMID 29260460
- See also: redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1692R00001&attachmentIdentifier=c4198b29-3cc2-4610-9434-d1ed7ba52643&fileName=D1692R00001_CSR_synopsis_redacted.pdf&versionIdentifier=